## Partnership Optimizes Weight Management in Primary Care (PROMISE) NCT02959021 February 3, 2022

## STATISTICAL ANALYSIS PLAN

To test the main hypotheses, longitudinal mixed effects models will be used to model the percent change in weight at 6, 12, and 18 months adjusted for baseline weight, using random effects to account for clustering within sites and the multiple observations per patient. The model will include time as categorical and use a group by time interaction to make best use of the data and to most precisely estimate temporal trends without assuming linearity. Differences in weight loss at each time point by study arm will be formally tested using estimated marginal means (also called LS-means).